CLINICAL TRIAL: NCT02944084
Title: Absorption and Excretion Kinetics of the Bioactive Ingredients of Rice Bran Extract
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: German Federal Ministry of Economics and Technology (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HS-RBE-2016
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Safety After Oral Intake; Pharmacokinetics After Oral Intake
Keywords: Bioavailability; Pharmacokinetics; Rice bran extract; Vitamin E; Gamma-oryzanol; Ferulic acid
MeSH Terms: interventions — Rice Bran Oil; Water; Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rice bran extract (Experimental): 2 g of unprocessed rice bran extract
  Interventions: Dietary Supplement: Rice bran extract
- Porridge in water (Experimental): 35 g of porridge containing 2 g of rice bran extract mixed with 95 ml of warm water
  Interventions: Dietary Supplement: Porridge in water
- Porridge in milk (Experimental): 35 g of porridge containing 2 g of rice bran extract mixed with 95 ml of warm milk (3.8% fat)
  Interventions: Dietary Supplement: Porridge in milk

INTERVENTIONS:
Dietary Supplement: Rice bran extract
  Arms: Rice bran extract
Dietary Supplement: Porridge in water
  Arms: Porridge in water
Dietary Supplement: Porridge in milk
  Arms: Porridge in milk

SUMMARY:
The oral absorption and urinary excretion kinetics of the bioactive ingredients from rice bran (gamma-oryzanol, tocotrienols, tocopherols and ferulic acid esters) after incorporation into an oat porridge (oat porridge) compared to unprocessed rice bran extract oil were investigated. The influence of the type of preparation (with water vs. milk) of porridge on the bioavailability of the bioactive compounds was compared. The study followed a single dose (2 g rice bran extract), randomized, three armed crossover study design with ≥1-week washout periods. Plasma and urine samples were collected at intervals up to 24 h after intake.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers with blood chemistry values within normal ranges

Age 18 to 35 years

BMI 19 to 25 kg per m2

Exclusion Criteria:

Pregnancy or lactation

Alcohol and or drug abuse

Use of dietary supplements or any medications except contraceptives

Any known malignant, metabolic and endocrine diseases

Previous cardiac infarction

Dementia

Participation in a clinical trial within the past 1 week prior to recruitment

Smoking

Physical activity of more than 5 h per wk

Lactose intolerance

Milk intolerance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve (AUC) of plasma concentration vs. time of total alfa, beta, gamma and delta tocopherols and tocotrienols [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
Mean area under the curve (AUC) of plasma concentration vs. time of total ferulic acid [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total ferulic acid after deconjugation with beta-glucuronidase/sulphatase
Mean area under the curve (AUC) of plasma concentration vs. time of total gamma-oryzanol [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
Mean maximum plasma concentration (Cmax) of total total alfa, beta, gamma and delta tocopherols and tocotrienols [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
Mean maximum plasma concentration (Cmax) of total ferulic acid [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total ferulic acid after deconjugation with beta-glucuronidase/sulphatase
Mean maximum plasma concentration (Cmax) of total gamma-oryzanol [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total gamma-oryzanol after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total alfa, beta, gamma and delta tocopherols and tocotrienols [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
Time to reach maximum plasma concentration (Tmax) of total ferulic acid [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total ferulic acid after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total gamma-oryzanol [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total gamma-oryzanol after deconjugation with beta-glucuronidase/sulphatase
Cumulative urinary excretion of total Vitamin E metabolites [nmol/g creatinine] | 0-24 h post dose
Cumulative urinary excretion of total ferulic acid [nmol/g creatinine] | 0-24 h post dose
Cumulative urinary excretion of total gamma-oryzanol [nmol/g creatinine] | 0-24 h post dose

SECONDARY OUTCOMES:
Serum aspartate transaminase activity [U/L] | 0, 4, 24h post-dose
Serum alanine transaminase activity [U/L] | 0, 4, 24h post-dose
Serum gamma-glutamyl transferase activity [U/L] | 0, 4, 24h post-dose
Serum alkaline phosphatase activity [U/L] | 0, 4, 24h post-dose
Serum bilirubin | 0, 4, 24h post-dose
Serum uric acid [mg/dL] | 0, 4, 24h post-dose
Serum creatinine [mg/dL] | 0, 4, 24h post-dose
Serum total cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum HDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum LDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum triacylglycerols [mg/dL] | 0, 4, 24h post-dose
LDL/HDL cholesterol ratio | 0, 4, 24h post-dose
Glomerular filtration rate [mL/min] | 0, 4, 24h post-dose
Serum glucose [mg/dL] | 0, 24h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Prof. Dr, Principal Investigator — University of Hohenheim
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Website of the research group — http://www.nutrition-research.de/